CLINICAL TRIAL: NCT03385330
Title: The Bronchopulmonary Dysplasia Saturation TARgeting (BPD STAR) Pilot Trial
Brief Title: BPD Saturation TARgeting
Acronym: BPD STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Sara B. DeMauro, MD MSCE, Assistant Professor of Pediatrics, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-014522
Record Dates: First submitted 2017-12-11; First posted 2017-12-28 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Bronchopulmonary Dysplasia; Chronic Lung Disease of Prematurity; Chronic Lung Disease
Keywords: BPD; Prematurity; Supplemental Oxygen; Oximetry; Infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LOWER oxygen saturation target group (Active Comparator): Oxygen saturation (SpO2) target range 90--94%. The study intervention will begin in the hospital and will continue at home until 6 months corrected age (CA). Overnight continuous oximetry will be transmitted wirelessly to the study team. In hospital, inspired oxygen will be adjusted as needed to maintain target SpO2. Monitoring will continue after discharge, and oxygen flow will be titrated monthly according to a standardized algorithm.
  Interventions: Other: LOWER oxygen saturation target group
- HIGHER oxygen saturation target group (Active Comparator): Oxygen saturation target range greater than or equal to 96%.The study intervention will begin in the hospital and will continue at home until 6 months CA. Overnight continuous oximetry will be transmitted wirelessly to the study team. In hospital, inspired oxygen will be adjusted as needed to maintain target SpO2. Monitoring will continue after discharge, and oxygen flow will be titrated monthly according to a standardized algorithm.
  Interventions: Other: HIGHER oxygen saturation target group

INTERVENTIONS:
Other: LOWER oxygen saturation target group — We will randomize infants with moderate or severe BPD to lower SpO2 target ranges. The study team will then use novel technology to monitor infants starting at randomization, continuing after discharge and until 6 months corrected age, titrating supplemental oxygen to achieve these target SpO2 ranges.
  Arms: LOWER oxygen saturation target group
Other: HIGHER oxygen saturation target group — We will randomize infants with moderate or severe BPD to higher SpO2 target ranges. The study team will then use novel technology to monitor infants starting at randomization, continuing after discharge and until 6 months corrected age, titrating supplemental oxygen to achieve these target SpO2 ranges.
  Arms: HIGHER oxygen saturation target group

SUMMARY:
Bronchopulmonary dysplasia (BPD), or chronic lung disease of prematurity, affects nearly half of extremely preterm infants.This study evaluates the use of supplemental oxygen to manage infants with established BPD. Participants will be randomly placed in either a higher oxygen saturation group or a lower oxygen saturation target group.

DETAILED DESCRIPTION:
Bronchopulmonary Dysplasia is diagnosed only in babies who are born prematurely, and affects about half of extremely preterm infants. The incidence of BPD has increased over time. It is most commonly defined as oxygen dependence at 36 weeks postmenstrual age (PMA).

Infants with BPD face more than doubled odds of death after 36 weeks PMA or disability at 5 years compared to preterm infants without BPD. BPD is associated with abnormal lung function throughout childhood and significantly increases health care costs. Cognitive and respiratory outcomes are closely linked throughout the life course; thus, optimal long--term management of BPD during infancy may ultimately improve cognitive outcomes of this high--risk population.

Supplemental oxygen is a lifesaving therapy for premature infants; yet, there is limited evidence about the safety or efficacy of using supplemental oxygen to target higher versus lower oxygen saturations in infants with established BPD.

Infants between the ages of 34-44 weeks post-menstrual age with moderate or severe BPD will be randomly assigned to higher or lower oxygen saturation target ranges. The study intervention will begin in the hospital and will continue at home until 6 months corrected age. When infants are discharged with supplemental oxygen, this will be titrated according to a study algorithm in order to ensure that the target saturations are maintained throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Pre-term males or females infants born at <30 0/7 weeks gestation at birth
* Current age 34 0/7 to 43 6/7 weeks postmenstrual age
* Diagnosis of moderate or severe Bronchopulmonary Dysplasia based on the NIH consensus definition
* Infant has never been discharged to home from the hospital

Exclusion Criteria:

* Congenital anomaly or oncologic process likely to affect growth or respiratory status
* Hemoglobinopathy or other blood disorder likely to affect oxygen saturations
* Contraindication to nasal cannula use (for example, severe nasal septal breakdown).
* Pulmonary hypertension requiring pharmacotherapy at the time of screening/enrollment.
* Tracheostomy
* Intubated during entire eligibility period

Ages: 34 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara DeMauro, MD, Principal Investigator — The Childrens Hospital of Pennsylvania
Locations (3):
- United States (3):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeMauro SB, Jensen EA, Passarella M, Gambacorta MC, Dhawan M, Weimer J, Jang S, Panitch H, Kirpalani H. Oxygen Saturation Targeting for Infants with Bronchopulmonary Dysplasia: A Pilot Randomized Trial. Ann Am Thorac Soc. 2025 Apr;22(4):560-569. doi: 10.1513/AnnalsATS.202404-443OC. PMID 40167293

RESULTS

PARTICIPANT FLOW:
Groups:
- LOWER Oxygen Saturation Target Group: Oxygen saturation target range 90--94%. The study intervention will begin in the hospital and will continue at home until 6 months CA. Overnight continuous oximetry will be transmitted wirelessly to the study team. In hospital, inspired oxygen will be adjusted as needed to maintain target SpO2. Monitoring will continue after discharge, and oxygen flow will be titrated monthly according to a standardized algorithm.
  LOWER oxygen saturation target group: We will randomize infants with moderate or severe BPD to lower SpO2 target ranges. The study team will then use novel technology to monitor infants starting at randomization, continuing after discharge and until 6 months corrected age, titrating supplemental oxygen to achieve these target SpO2 ranges.
Period: Overall Study
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Started | 28 | 22
Completed | 23 | 19
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group | Total
Number analyzed (Participants) | 28 | 22 | 50
Age, Continuous [Mean (Standard Deviation); unit: post-menstrual age (PMA) in weeks] — Postmenstrual age (PMA) at enrollment
  post-menstrual age (PMA) in weeks | 39.9 (2.3) | 40.5 (2.2) | 40.2 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 25 | 20 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 15 | 34
  White | 7 | 5 | 12
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intermittent Hypoxemia (IH) Events Per 8 Hours of Monitoring Time
Description: Incidence of intermittent hypoxia (IH, defined as SpO2 <80% for >=30 seconds), reported as median number of events per 8 hours of monitoring time.
Time Frame: Between discharge and 6 months corrected age
Population: Infants with sufficient oximetry data were included in primary outcome analyses.
Measure: Median (Inter-Quartile Range); unit: IH events per 8 hours of monitoring time
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Number analyzed (Participants) | 25 | 19
IH events per 8 hours of monitoring time | 2.2 [1.0 to 4.2] | 1.2 [0.3 to 3.1]

2. Secondary Outcome: Duration of Hypoxia - Proportion of Monitored Time With Oxygen Saturation <80%
Description: Total exposure to hypoxia - proportion of monitored time with SpO2 <80%
Time Frame: Between discharge and 6 months corrected age
Population: Analysis includes infant with sufficient oximetry data
Measure: Median (Inter-Quartile Range); unit: proportion of monitored time
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Number analyzed (Participants) | 25 | 19
proportion of monitored time | 0.005 [0.001 to 0.016] | 0.004 [0.001 to 0.013]

3. Secondary Outcome: Change in Weight Z-score
Description: Change in weight Z-score. A Z-score of 0 represents average weight. Positive change in Z score indicates increasing weight relative to the population average weight. Negative change in Z score indicates decreasing weight relative to the population average weight.
Time Frame: Between randomization and 6 months corrected age
Measure: Mean (Standard Deviation); unit: delta Z-score
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Number analyzed (Participants) | 27 | 22
delta Z-score | 0.6 (1.4) | 0.5 (1.2)

4. Secondary Outcome: Change in Length Z-score
Description: Change in length Z-score. A Z-score of 0 represents average length. Positive change in Z score indicates increasing length relative to the population average length. Negative change in Z score indicates decreasing length relative to the population average length.
Time Frame: Between randomization and 6 months corrected age
Measure: Mean (Standard Deviation); unit: delta Z-score
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Number analyzed (Participants) | 27 | 22
delta Z-score | 1.7 (1.3) | 1.2 (1.4)

5. Secondary Outcome: Change in Head Circumference Z-score
Description: Change in head circumference (HC) Z-score. A Z-score of 0 represents average HC. Positive change in Z score indicates increasing HC relative to the population average HC. Negative change in Z score indicates decreasing HC relative to the population average HC.
Time Frame: Between randomization and 6 months corrected age
Measure: Mean (Standard Deviation); unit: delta Z-score
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Number analyzed (Participants) | 27 | 22
delta Z-score | 0.5 (1.3) | 0.4 (1.7)

6. Secondary Outcome: Number of Participants With Re-hospitalization
Description: Any re-hospitalization
Time Frame: Between discharge and 6 months corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Number analyzed (Participants) | 28 | 22
Participants | 9 | 6

7. Secondary Outcome: Number of Participants With Respiratory Medication Use
Description: Number of patients with inhaled respiratory medication use
Time Frame: At 6 months corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Number analyzed (Participants) | 28 | 22
Participants | 6 | 6

8. Secondary Outcome: Number of Participants With Visits to Emergency Room or Urgent Care for Respiratory Reasons
Description: Any visits to ER or urgent care for respiratory health-related problems
Time Frame: Between discharge and 6 months corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Number analyzed (Participants) | 28 | 22
Participants | 5 | 2

9. Secondary Outcome: Feeding
Description: Quality of infant oral feeding skills, parent reports that the child's feeding times are stressful or very stressful for themselves
Time Frame: At 6 months corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Number analyzed (Participants) | 21 | 15
Participants | 1 | 0

10. Secondary Outcome: Development
Description: Bayley Scales of Infant Development screening test, which is a standardized assessment of cognitive, motor, and language development in infancy and early childhood. Outcome will be reported as number of children considered "at risk" in any domain.
Time Frame: At 6 months corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
Number analyzed (Participants) | 23 | 19
Participants | 8 | 3

ADVERSE EVENTS:
Time Frame: Data were collected between enrollment and 6 months corrected age
Arm/Group | LOWER Oxygen Saturation Target Group | HIGHER Oxygen Saturation Target Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/22
Other Adverse Events (participants affected / at risk) | 0/28 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03385330/Prot_SAP_002.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT03385330/ICF_003.pdf